CLINICAL TRIAL: NCT05918497
Title: Comparison Between Variable Time Regimen of Dosing L-Thyroxine for Treatment Hypothyroid Fasting Ramadan
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Ahmed Mohamed, lecturer of internal medicine, Sohag University
Other Study IDs: Soh-Med-23-04-08PD.
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-04

CONDITIONS: Different Regimens in Treatment of Hypothyroidism During Fasting in Ramadan
Keywords: levothyroxin , hypothyroidism , fasting in Ramadan
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: .patients who will switch to twice weekly dosing. Their weekly dose was divided equally into those doses, given at successive fixed days of the week
- Group 2: patients who will switch to once-weekly dosing.
- Group 3: patients who will continue to take L T4 on a standard daily basis.

SUMMARY:
This is a study aiming to report the effect of a variable time regimen of L T4 during Ramadan, as an easier alternative, on adherence and thyroid status after Ramadan compared to standard daily dosing.

DETAILED DESCRIPTION:
Patient and Method This a prospective study will be including Muslim hypothyroid patients willing to fast Ramadan during the year 2023 attending outpatient clinic, Sohag faculty of medicine, Sohag university, Egypt.

All included patients will be euthyroid, and stable on the same L T4 dose for at least 3 months before the start of Ramadan.

Exclusion criteria will be thyroid cancer patients requiring suppressive therapy, central hypothyroidism, pregnancy, coronary heart disease, arrythmia, chronic heart failure, liver cirrhosis, renal failure, acute medical, or surgical illness at the time of evaluation to avoid acute and chronic non thyroidal illness syndromes.

the patients will be divided into three groups. Group 1 patients who will switch to twice weekly dosing. Their weekly dose was divided equally into those doses, given at successive fixed days of the week. Group 2 patients who will switch to once weekly dosing. Group 3 patients who will continue to take L T4 on standard daily basis.

Patients from are free to follow one of four L T4 regimens during Ramadan, regimen 1: to take L T4 60 min before Iftar and beverages, regimen 2: to take L T4 3-4 h after Iftar, 60 min before Suhor meal, regimen 3: to take L T4 before the start of next fast 3 4 h after an early Suhor at midnight. If patients mixed between regimens 1 and 2, this was labeled regimen 4.

Adherence will assess by interviewing participants during post Ramadan visit. Nonadherence define as stopping food and beverages for less than 3 h before L T4 tablet(s) or stopping food and beverages for less than 45 min after L T4 tablet(s). Patients who skipped L T4 treatment for 2 or more days without making up for their missed doses will be excluded from the study.

Thyroid status will reassess in post Ramadan visit using TSH, provided that this visit comes within 6 weeks from the end of Ramadan.

Ethical aspect Informed written consent will be taken from all patients to include their data in the study. The research will be approved by medical ethics committee of Sohag University Faculty of Medicine Statistical analysis Data will be analyzed using STATA version 14.2 (Statistical Software: Release 14.2 College Station, TX: Stata Corp LP). Quantitative data will be represented as mean, standard deviation, median and range. normally distributed. Qualitative data will be presented as numbers and percentages. Chi square test will be used for comparison of percentages in different groups. P value will be considered significant if it was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

- All included patients will be euthyroid, and stable on the same L T4 dose for at least 3 months before the start of Ramadan.

Exclusion Criteria:

* Exclusion criteria will be thyroid cancer patients requiring suppressive therapy, central hypothyroidism, pregnancy, coronary heart disease, arrythmia, chronic heart failure, liver cirrhosis, renal failure, acute medical, or surgical illness at the time of evaluation to avoid acute and chronic non thyroidal illness syndromes.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: including Muslim hypothyroid patients willing to fast Ramadan during the year 2023 attending outpatient clinic, Sohag faculty of medicine, Sohag university, Egypt
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison Between Variable Time Regimen of Dosing L-Thyroxine for Treatment Hypothyroid Fasting Ramadan | 2 months after ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kasem, lecturer, Study Chair — sohag university .faculty of medicine; Ahmed Faysal, lecturer, Study Chair — sohag university .faculty of medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided